CLINICAL TRIAL: NCT06906432
Title: Multimodal Omics and Imaging Study on the Mechanisms of Brain-heart Injury in Patients With Intracranial Hemorrhage
Brief Title: Mechanisms of Brain-Heart Injury of Post-Intracranial Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Youyi Hospital (Unknown); Tianjin Medical University General Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Gulou Hospital Affiliated to Medical College of Nanjing University (Unknown)
Responsible Party: Principal Investigator, Dr. Yong Cao, Dr., Beijing Tiantan Hospital
Other Study IDs: BHI2024
Record Dates: First submitted 2025-02-11; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Cerebrocardiac Syndrome; Mass Spectrometry; Heart Failure; Atrial Fibrillation; Ischemic Heart Disease; Heart Infarction; Arrhythmias, Cardiac; Delayed Cerebral Ischemia; Hydrocephalus; Vasospasm, Cerebral; Intracerebral Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Neurocirculatory Asthenia; Heart Failure; Atrial Fibrillation; Myocardial Ischemia; Myocardial Infarction; Arrhythmias, Cardiac; Hydrocephalus; Vasospasm, Intracranial; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and cerebrospinal fluid (CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with intracranial hemorrhage: patients with subarachnoid hemorrhage or intracerebral hemorrhage
  Interventions: Diagnostic Test: Multi-disciplinary assessment

INTERVENTIONS:
Diagnostic Test: Multi-disciplinary assessment — Multi-disciplinary assessment including blood tests, CSF test, electrocardiograms, ultrasound, imaging, etc

SUMMARY:
Intracranial hemorrhage is a condition characterized by high mortality rates and suboptimal functional outcomes. It precipitates both direct brain injury and subsequent secondary injuries, including delayed cerebral ischemia, brain edema, and hydrocephalus. Complications such as cardiac injury may also arise, categorizing them within the cerebrocardiac syndrome (CCS). The clinical spectrum of CCS encompasses acute myocardial injury, acute coronary syndrome, left ventricular systolic and diastolic dysfunction, cardiac arrhythmias, and sudden cardiac death, all of which are associated with increased mortality and deterioration in patient status. The precise pathophysiological mechanisms underlying both cerebral and cardiac injuries remain enigmatic, and the implications for diagnosis and therapeutic strategies are yet to be fully explored.

In this study, we propose to enroll patients with intracranial hemorrhage who will undergo conventional treatment and comprehensive multidisciplinary evaluations. Our observational research is grounded in a multimodal omics and imaging approach, aimed at investigating both local and systemic injuries subsequent to intracranial hemorrhage. This comprehensive strategy is intended to facilitate precise diagnosis, risk stratification, and clinical decision-making, while also shedding light on the pathophysiological mechanisms involved.

The primary objectives of this research are to address the following key questions:

* [Question 1] What are the pathophysiological mechanisms underlying cardiac injury in patients with intracranial hemorrhage?
* [Question 2] What are the pathophysiological mechanisms responsible for early and delayed brain injuries following intracranial hemorrhage?"

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older at the time of enrollment.
2. Acute intracranial hemorrhage confirmed by neuroimaging (CT, MRI，CTA, MRA, or DSA) within 48 hours of symptom onset.
3. Ability to provide informed consent or have a legally authorized representative willing to consent on their behalf.

Exclusion Criteria:

1. Patients who refuse to participate in the study or cannot provide informed consent.
2. Patients with a history of significant cardiovascular disease, including myocardial infarction, heart failure, or arrhythmias, unless stable and well-controlled.
3. Patients who have undergone cardiac bypass surgery, stent placement, or other cardiovascular interventions within the past 6 months.
4. Patients with active brain tumors, ischemic stroke within 3 months or a history of previous brain injury that could confound the study findings.
5. Patients with active malignant disease, severe inflammatory or infectious disease, or those who have undergone surgery for any reason within the past 3 months.
6. Patients with any condition that, in the opinion of the investigator, would make it unsafe or impractical to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we intend to enroll patients suffering from acute intracranial hemorrhage, who will undergo both conventional therapy and comprehensive multidisciplinary evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2034-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Short-term cardiac events | At discharge (assessed up to 5 days)
  Participants who suffer from sudden dysfunction or structural abnormalities of the heart (e.g., arrhythmias, myocardial infarct, sudden death) confirmed through:
  1. Electrocardiogram (ECG);
  2. Cardiac biomarkers (e.g., troponin);
  3. Echocardiography;
  4. Holter monitoring.
Long-term cardiac events | 3 months post-discharge
  Participants who suffer from sudden dysfunction or structural abnormalities of the heart (e.g., arrhythmias, myocardial infarct, sudden death) confirmed through:
  1. Electrocardiogram (ECG);
  2. Cardiac biomarkers (e.g., troponin);
  3. Echocardiography;
  4. Holter monitoring.
Short-term delayed cerebral ischemia | At discharge (assessed up to 5 days)
  Participants who suffer from secondary reduction in cerebral blood flow due to mechanisms such as vasospasm, microthrombosis, or hemodynamic disturbances, confirmed through:
  1. Head CT/MRI;
  2. Transcranial doppler sonography (TCD).
Long-term delayed cerebral ishemia | 3 months post-discharge
  Participants who suffer from secondary reduction in cerebral blood flow due to mechanisms such as vasospasm, microthrombosis, or hemodynamic disturbances, confirmed through:
  1. Head CT/MRI;
  2. Transcranial doppler sonography (TCD).
Short-term brain-heart syndrome | At discharge (assessed up to 5 days)
  Participants who suffer from cardiac dyafunction triggered by cerebral hemorrhage. Clinical manifestations include ECG abnormalities (ST-T changes, prolonged QT interval, arrhythmias), elevated cardiac enzymes (e.g., troponin), cardiac insufficiency (e.g., heart failure, pulmonary edema), chest pain mimicking myocardial ischemia and myocardial infarct. Some patients may develop life-threatening arrhythmias (e.g., ventricular fibrillation). Diagnostic evaluations involve:
  1. Electrocardiogram (ECG);
  2. Cardiac enzyme tests (e.g., troponin, CK-MB);
  3. Echocardiography;
  4. Brain imaging (CT/MRI);
  5. Biomarkers (e.g., BNP).
Long-term brain-heart syndrome | 3 months post-discharge
  Participants who suffer from cardiac dyafunction triggered by cerebral hemorrhage. Clinical manifestations include ECG abnormalities (ST-T changes, prolonged QT interval, arrhythmias), elevated cardiac enzymes (e.g., troponin), cardiac insufficiency (e.g., heart failure, pulmonary edema), chest pain mimicking myocardial ischemia and myocardial infarct. Some patients may develop life-threatening arrhythmias (e.g., ventricular fibrillation). Diagnostic evaluations involve:
  1. Electrocardiogram (ECG);
  2. Cardiac enzyme tests (e.g., troponin, CK-MB);
  3. Echocardiography;
  4. Brain imaging (CT/MRI);
  5. Biomarkers (e.g., BNP).

SECONDARY OUTCOMES:
Short-term modified Rankin Scale scores | At discharge (assessed up to 5 days)
  The modified Rankin Scale (mRS) scores of participants evaluated by specialists. The mRS scores range form 0 to 6, with higher scores indicating worse outcomes.
Long-term modified Rankin Scale scores | 3 months post-discharge
  The modified Rankin Scale (mRS) scores of participants evaluated by specialists. The mRS scores range form 0 to 6, with higher scores indicating worse outcomes.

OTHER OUTCOMES:
Lower extremity deep venous thrombosis | At discharge (assessed up to 5 days)
  Participants who suffer from lower extremity deep venous thrombosis confirmed by lower vein ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No